CLINICAL TRIAL: NCT04959292
Title: Meniscus Regeneration After Meniscectomy: Factors Predicting the Regeneration and the Clinical Significance of the Regenerated Meniscus
Brief Title: Meniscus Regeneration After Meniscectomy and Its Clinical Significance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019299
Record Dates: First submitted 2021-06-16; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Meniscus Rupture; Regeneration
Keywords: meniscus; regeneration; meniscectomy
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — resected meniscus and biopsy of regenerated meniscus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meniscus regeneration: Reconstruction of the anterior cruciate ligament, total or partial meniscus resection was performed in our hospital, and two years after the operation, the meniscus regeneration was found under secondary arthroscopy.
  Interventions: Diagnostic Test: arthroscopy
- Meniscus without regeneration: Anterior cruciate ligament reconstruction, total or partial meniscus resection was performed in our hospital, and two years after the operation, no meniscus regeneration was found under secondary arthroscopy.
  Interventions: Diagnostic Test: arthroscopy

INTERVENTIONS:
Diagnostic Test: arthroscopy — arthroscopy

SUMMARY:
Meniscus injury is common in sports-active population, and partial or total meniscectomy is standard surgery for meniscal tear. Meniscus plays an important role in load transferring, shock absorbing, knee joint stabilizing and chondral protection. Plenty of studies indicate that meniscus-deficiency increases the risk of OA and cause long-term poor outcomes.

Spontaneous human meniscus regeneration is rarely reported and whether regenerated meniscus is chondral-protective and can prevent OA progression remain unknown. During our clinical practice, we have encountered many cases with complete meniscal regeneration under arthroscopy. In this study, we will include all the patients who receiving meniscectomy and ACL reconstruction and knee arthroscopy 2 years after primary surgery. Patients demographic characters will be reviewed. The resected meniscus in the primary surgery and biopsied regenerated meniscus will be analyzed by histological and immunohistochemical method and their ultrastructure will be observed by electron microscope. Patients will be followed at 2-, 5- and 10-year after the primary surgery and the cartilage degeneration and OA progression will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients intending to undergo single-knee ACL reconstruction at our Institute of Sports Medicine.
2. The age of 18 ~ 50 years old at the time of operation.
3. Both men and women.
4. BMI < 24.
5. Complete or partial meniscectomy was performed at the same time as ACL reconstruction.
6. Patients willing to undergo a second arthroscopic exploration 2 years postoperatively and to take the portal screws used to fix the ligaments during the initial surgery.
7. Patients with preserved meniscus video during ACL reconstruction.
8. The degree of knee osteoarthritis (KOA) at the time of operation was < Ⅲ of Kellgren Laurence level.

Exclusion Criteria:

1. Patients with severe knee cartilage injury.
2. Patients with KOA≥KLⅢ at the time of operation.
3. The patients cannot be followed up.
4. Patients who refused the second arthroscopy and the removal of the internal fixation portal screw at the time of surgery.
5. Patients with rheumatoid arthritis or other arthritis.
6. Patients with other systemic diseases who take oral anti-inflammatory analgesics for years.
7. Patients with multiple injections of drugs in the joint due to various reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all the patients receving meniscectomy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
meniscus regeneration | 2 year
  the resected meniscus regeneration is found under the arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Zimu Mao, Dortor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No